CLINICAL TRIAL: NCT06695780
Title: Exploration Des Typologies Alimentaires Et Caractérisation Par Un Phénotypage Multidimensionnel D'une Population De Personnes Âgées De La Région Auvergne-Rhône Alpes
Brief Title: Food Typologies and Multidimensional Phenotyping of Elderly in Auvergne-Rhône-Alpes (Part'AGE)
Acronym: Part'AGE
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Icadom (Industry); Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-AO1319-38
Record Dates: First submitted 2024-11-18; First posted 2024-11-19 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Nutritional Assessment; Physical Activity; Health; Oral Health
Keywords: eating behaviors; elderly; health; phenotyping; food typologies; prevention
MeSH Terms: conditions — Motor Activity; Feeding Behavior | interventions — Exercise; Health Status

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dried whole blood; Urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: survey on eating behavior, physical activity and health status — Participatory research: participants will carry out surveys, functional tests and urine and blood sampling completely independently

SUMMARY:
To better understand how diet influences health during aging, the French National Research Institute for Agriculture, Food and the Environment (INRAE) is working with the Gérontopôle Auvergne-Rhône-Alpes on a project called Part'AGE. Part'AGE is a participatory research project where researchers want to recruit 1,000 people aged between 55 and 75 years, men and women, living in Auvergne-Rhône-Alpes in urban or rural areas. The goal is to study eating habits and state of health. To do this, researchers will examine many factors that can influence them, such as physical activity, overall health, consumption patterns or territories. Researchers will collect detailed information to classify participants into different groups (food typologies) based on their eating habits and state of health. With this distribution, the goal is to be able to give each group personalized nutritional advice to age in better health.

To participate in the study, the participants will need to collect a few drops of blood from the end of the finger, a urine sample, and do some tests (mobility, oral health). It will also be necessary to fill out questionnaires on eating habits, physical activity, and other aspects that may influence health. The benefices for to participants will be to contribute to nutrition research and to receive personalized feedback and advices on eating habits.

DETAILED DESCRIPTION:
The main objective of the study is to characterize the food consumption profile of a population of people aged 55 to 75, men and women, living in the Auvergne-Rhône-Alpes region, either in an urban or rural environment. The aim is to classify volunteers into dietary typologies associated with more or less successful aging. Thus, the investigators will classify volunteers into five dietary typologies:

1. Typology "at risk of malnutrition": volunteers who do not cover their daily protein-energy needs, i.e. having daily protein-energy intakes estimated by food consumption data lower than the needs estimated by the Mifflin and St Jeor equation (based on anthropometric and physical activity measurements).
2. "Balanced diet without cardio-metabolic risk" typology: volunteers covering their daily protein-energy needs, with an aHEI (Alternative Healthy Eating Index) score greater than 80 and with a waist circumference less than or equal to 94 cm for men and 80 cm for women.
3. "Diet to improve without cardio-metabolic risk" typology: volunteers covering their daily protein-energy needs, with an aHEI score less than or equal to 80 and with a waist circumference less than or equal to 94 cm for men and 80 cm for women.
4. "Balanced diet with cardio-metabolic risk" typology: volunteers covering their daily protein-energy needs, with an aHEI score greater than 80 and with a waist circumference greater than 94 cm for men and 80 cm for women.
5. Typology "diet to improve with cardio-metabolic risk": volunteers covering their daily protein-energy needs, presenting an aHEI score less than or equal to 80 and with a waist circumference greater than 94 cm for men and 80 cm for women.

For each of these dietary typologies, the investigators will explore the diversity of: cardio-metabolic capacities; diet; mobility; health status (oral health, intestinal health, stress, fatigue, anxiety, sleep, addictions); the psychological-socio-economic dimension; biological parameters obtained after the collection of biological samples.

This study will be entirely carried out by correspondence, without the volunteers needing to travel. Wide communication on the study will first be carried out in Auvergne-Rhône-Alpes. A phone number and an email address of the research team will be left for people wishing more information. Volunteers will directly contact the administrative agent in charge of selection in order to leave their contact details. The administrative agent will respond or contact the participants in return to present the study in its entirety, tell them about their rights, and check their eligibility. If they are eligible and interested, volunteers will be sent the information form and a connection guide by email or by post and an appointment will be scheduled for a dematerialized inclusion visit with a study investigator. The inclusion visit will be carried out remotely, from a secure platform. Upon receipt of consent, the investigators will assign an identification number to the volunteer and will trigger the sending by post of a phenotyping BOX to their home containing all the material necessary to carry out the study, accompanied by an explanatory note. The volunteers will connect to a secure platform to complete 29 questionnaires, will carry out functional tests and anthropometric measurements and will collect their biological samples (blood drops and urine). Volunteers will send their biological samples to the INRAE laboratory within 2 days of their collection.

In return, volunteers will have the opportunity to:

* participate in the regional hubs of the Part'AGE project: these hubs will be made up of nutrition-prevention-health stakeholders for successful aging. The trial volunteers will thus be able to participate in the collective meetings of these hubs to benefit from overall feedback on the project and awareness of the different dimensions studied within the framework of the protocol.
* Personalized feedback proposed by the investigator at the end of the project, including a qualitative assessment of dietary typology of participants, as well as their strengths and weaknesses on the other dimensions studied. This assessment will provide an image of their own typology, but also provide a benchmark in relation to other volunteers (averages), also depending on the territories.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (balanced sex ratio or at least 40% male to 60% female) in complete autonomy at home.
* 55 to 75 years old, including the limits
* 20 ≤ BMI ≤35 kg/m2
* Available to carry out the entire protocol, including self-sampling (not sensitive to the sight of one's own blood for example) and agreeing to stop taking food supplements during the study.
* Having a scale available: at home, pharmacy, family, etc.
* Having internet access and a device with a screen and camera (PC, tablet, smartphone, etc.) at home or able to go to a project partner (CCAS, Point France Service, Community, Association, etc.) that can provide this access
* Subject agreeing to give written consent (by phone or videoconferencing), and registration in the national file of volunteers who participate in research
* Person declaring to be subject to a social security scheme.

Exclusion Criteria:

* Weight loss ≥ 5% in 1 month or ≥ 10% in 6 months or ≥ 10% compared to usual weight
* Treated diabetes
* Sub-acute pathology (flu, gastroenteritis, bacterial infection, etc.) or trauma (fracture, surgical intervention, etc.) in the 30 days prior to inclusion.
* Hepatocellular insufficiency,
* Heart failure with decompensation,
* Renal insufficiency (clearance <30 ml/min)
* Chronic anti-inflammatory treatment, long-term corticosteroid therapy > 1 month, infiltration
* Progressive pathology at the time of inclusion (cancer, etc.)
* Gastrointestinal pathology deemed incompatible with the protocol
* Unstable thyroid diseases
* Recent change in eating habits in the last 30 days (weight loss diet, veganism, intermittent fasting, ketogenic diet, etc.)
* Intense physical activity (activity causing shortness of breath and sweating) > 10 hours per week
* Person in a period of exclusion from the National File of Healthy Volunteers
* Subject under guardianship, curator-ship, deprived of liberty or under judicial protection

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Auvergne-Rhône-Alpes region, taking care to recruit both urban and rural people.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Classification of our study population into 5 dietary typologies associated with more or less successful aging | From enrollment to the end of the surveys at 30 days
  1. Typology "at risk of malnutrition": volunteers who do not cover their daily protein-energy needs, i.e. having daily protein-energy intakes estimated by food consumption data lower than the needs estimated by the Mifflin and St Jeor equation (based on anthropometric and physical activity measurements).
  2. "Balanced diet without cardio-metabolic risk" typology: volunteers covering their daily protein-energy needs, with an aHEI (Alternative Healthy Eating Index) score greater than 80 and with a waist circumference less than or equal to 94 cm for men and 80 cm for women.
  3. "Diet to improve without cardio-metabolic risk" typology: volunteers covering their daily protein-energy needs, with an aHEI score less than or equal to 80 and with a waist circumference less than or equal to 94 cm for men and 80 cm for women.
  4. "Balanced diet with cardio-metabolic risk" typology: volunteers covering their daily protein-energy needs, with an aHEI score greater than 80 and with a waist circumference

SECONDARY OUTCOMES:
Blood parameters and waist-to-hip ratio | From enrollment to the end of the surveys at 30 day
  Assessment of glucose, C-peptide, triglycerides, cholesterol, amino acids, prealbumin and CRP levels in fingertip blood collected at home, and waist-to-hip ratio.
Assessment of dietary habits and choices | From enrollment to the end of the surveys at 30 day
  Assessment of dietary habits and choices by: polyphenol-targeted food frequency questionnaire, appetite questionnaire (Council on Nutrition Appetite Questionnaire, CNAQ), questionnaire on food expectations and choices, on culinary practices, supply, and nutritional perceptions. Assessment of diet quality with various scores (DQI, PNNS-GS, DII) and post-hoc analyses.
Assessment of physical capacities and physical activity | From enrollment to the end of the surveys at 30 day
  Assessment of physical capacities and physical activity with the chair rise test, calf circumference measurement and two questionnaires (IPAQ, and RPAQ/ONAPS) aimed at assessing physical activity and sedentary lifestyle.
Assessment of several dimensions of health | From enrollment to the end of the surveys at 30 day
  Assessment of several dimensions of health: 1) oral health (masticatory performance, number of posterior functional units, GOHAI questionnaire on quality of life related to oral health, EAT-10 questionnaire on dysphagia/swallowing, XI questionnaire on dry mouth and the CIF questionnaire on oral dysfunctions); 2) intestinal health (intestinal transit questionnaire and intestinal comfort questionnaire (IGQ); 3) various aspects of quality of life (stress, fatigue, anxiety, sleep, addictions, etc.).
Assessment of psycho-socio-economic status | From enrollment to the end of the surveys at 30 day
  Assessment of psycho-socio-economic status: questionnaire on precariousness (EPICES score), loneliness (De Jong Gierveld scale), desired healthy aging, quality of life (CAPS-19 scale), well-being profile, satisfaction and frustration of basic psychological needs. Assessment of personality traits and budget dedicated to food purchases.
Collection of blood and urine samples. | From enrollment to the end of the surveys at 30 day
  Collection of blood and urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Lahaye, MD, Ph D, Study Chair — Unité mobile de Gériatrie - Centre Hospitalier Universitaire- Site Gabriel Montpied
Locations (2):
- France (2):
  - ICADOM, Meylan, Isere
  - Centre de Recherche en Nutrition Humaine Rhône-Alpes, Pierre-Bénite, Rhone

IPD SHARING:
Plan to Share IPD: No
As soon as possible, results will be published. Upon requests, sharing of data could be considered on a case-by-case basis.

REFERENCES:
- [Background] de Toro-Martin J, Arsenault BJ, Despres JP, Vohl MC. Precision Nutrition: A Review of Personalized Nutritional Approaches for the Prevention and Management of Metabolic Syndrome. Nutrients. 2017 Aug 22;9(8):913. doi: 10.3390/nu9080913. PMID 28829397
- [Background] Berry SE, Valdes AM, Drew DA, Asnicar F, Mazidi M, Wolf J, Capdevila J, Hadjigeorgiou G, Davies R, Al Khatib H, Bonnett C, Ganesh S, Bakker E, Hart D, Mangino M, Merino J, Linenberg I, Wyatt P, Ordovas JM, Gardner CD, Delahanty LM, Chan AT, Segata N, Franks PW, Spector TD. Human postprandial responses to food and potential for precision nutrition. Nat Med. 2020 Jun;26(6):964-973. doi: 10.1038/s41591-020-0934-0. Epub 2020 Jun 11. PMID 32528151
- See also: Project web site — https://www.tetrae.fr/les-projets/partage